CLINICAL TRIAL: NCT00711620
Title: Multicenter, Randomized, Controlled Study to Evaluate the Efficacy of Thymosin alpha1 in Patients With Severe Sepsis
Brief Title: Efficacy of Thymosin alpha1 for Severe Sepsis
Acronym: ETASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Guan Xiangdong, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007015
Record Dates: First submitted 2008-06-27; First posted 2008-07-09 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2009-10

CONDITIONS: Severe Sepsis
Keywords: sepsis; Immunotherapy; Thymosin
MeSH Terms: conditions — Sepsis | interventions — Thymalfasin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thymosin alpha 1+Standard Therapy (Experimental): Patients receive treatment based on SSC guideline with additional thymosin alpha1
  Interventions: Drug: Thymosin alpha 1
- normal saline+standard therapy (Placebo Comparator): Patients receive treatment based on SSC guideline with additional normal saline.
  Interventions: Drug: Thymosin alpha 1

INTERVENTIONS:
Drug: Thymosin alpha 1 — 1.6 mg s.c injection twice per day for 5 days, then 1.6 mg s.c injection once per day for 2 days.
  Other Names: Zadaxin

SUMMARY:
The purpose of this study is to evaluate the efficacy of thymosin alpha 1 for treating severe sepsis.

DETAILED DESCRIPTION:
Severe sepsis is a disease of infectious origin with a high risk of death. Over the past decade, thymosin alpha1 have already provided clinicians with additional weapon in the fight against infectious diseases, but it is unknown whether thymosin alpha1 is effective in treating severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis according to ACCP/CCM criteria
* Patient or legally authorized representative able to provide informed consent

Exclusion Criteria:

* Subject is less than 18 years or more than 85 years of age
* If female, the subject is pregnant or nursing
* Subject is receiving immunosuppressive therapy such as cyclosporine, azothioprine,or cancer-related chemotherapy
* Patient not expected to survive 28 days because of uncorrectable medical condition, such as poorly controlled neoplasm or other end-stage disease
* History of bone marrow, lung, liver, pancreas, or small-bowel transplantation
* Acute pancreatitis with no established source of infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
28-day Mortality | 28 days
  The prospectively defined primary end point was death from any cause and was assessed 28 days after the start of the infusion.

SECONDARY OUTCOMES:
SOFA score | 7 days
  SOFA score was measured on day0, 3 and 7 after the start of the infusion in both groups.
Immune response to Thymosin alpha 1 | 7 days
  HLA-DR expression on CD14+,ratio between CD4+ and CD8+, CRP on day 0, 3, 7 after the start of the infusion in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Guan Xiangdong, M.D, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wu J, Zhou L, Liu J, Ma G, Kou Q, He Z, Chen J, Ou-Yang B, Chen M, Li Y, Wu X, Gu B, Chen L, Zou Z, Qiang X, Chen Y, Lin A, Zhang G, Guan X. The efficacy of thymosin alpha 1 for severe sepsis (ETASS): a multicenter, single-blind, randomized and controlled trial. Crit Care. 2013 Jan 17;17(1):R8. doi: 10.1186/cc11932. PMID 23327199